CLINICAL TRIAL: NCT05926843
Title: Evaluation of Spinal Cord Stimulation Assisted by Motor Rehabilitation Training for Restoring Motor Function After Spinal Cord Injury: an Interventional, Prospective, Monocentric Study
Brief Title: Spinal Cord Stimulation Assisted by Motor Rehabilitation Training for Restoring Motor Function After Spinal Cord Injury
Acronym: NeuroSCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Principal Investigator, Albano Luigi, MD, PhD, Assistant Professor of Neurosurgery, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neuro-SCS-001
Record Dates: First submitted 2023-06-01; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Spinal Cord Injuries
Keywords: motor restoration; chronic pain; rehabilitation; neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with functionally complete/incomplete spinal cord injury (Experimental): Individuals with functionally complete/incomplete spinal cord injury (ASIA grade A, B or C) who will undergo SCS for chronic pain
  Interventions: Procedure: Spinal cord stimulation surgery (device) and motor rehabilitation

INTERVENTIONS:
Procedure: Spinal cord stimulation surgery (device) and motor rehabilitation — The first part of the study will involve a preoperative evaluation. Participants' clinical history, neurological, neurophysiological and advanced brain/spine MRI examination will be assessed (Part 1). Subsequently, participants will undergo spinal cord stimulation surgery which involves the implantation of a medical device (Part 2). After the surgery, the research participants will be hospitalized at the Neurosurgery Unit (10 days) to monitor the incision site (Part 3). Thereafter, the patients will be moved (for at least 6 weeks) to the Rehabilitation Unit in order to identify appropriate stimulation parameters for inducing stepping and standing and for starting training. The combination of epidural stimulation with manual step/stand training will be thus evaluated (Part 4). Patients will be finally assessed by clinical evaluation, advanced MRI and neurophysiological examination to study the brain, spine and peripheral functions after six months (Part 5).

SUMMARY:
Interventional prospective longitudinal on the evaluation of spinal cord stimulation (SCS) assisted by motor rehabilitation training for restoring motor function in patients with spinal cord injury (SCI). The investigators will enroll ten research participants with clinically incomplete/complete SCI (patients with paraplegia or severe paraparesis) who will undergo SCS subsequently assisted by motor rehabilitation training for restoring motor function at IRCCS Ospedale San Raffaele, Milan, Italy. The main goal of the project is to evaluate the improvement in motor function generated by the combination of SCS and locomotor training. In line with recently published studies, the investigators propose that daily locomotor training in the presence of SCS with continuous stimulation parameters setting will enable the SCI individuals to stand and step independently while bearing full weight.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCI from at least one-year post injury;
* Complete or incomplete spinal cord damage (ASIA grade A, B or C) conditioning chronic neuropathic pain and motor impairment
* Age > 18 years;
* Indication to spinal cord stimulation surgery for chronic pain;
* Be unable to stand or step independently;
* No current anti-spasticity medication regimen;
* No botox injections in the prior 3 months;
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study;
* Willingness and ability to comply with scheduled visits and other trial procedures.

Exclusion Criteria:

* Any person unable to lie still within the environment of the MRI scanner for the required period to perform the study and those where MRI scanning is contraindicated (i.e. metal clips, claustrophobia);
* Pregnancy or breastfeeding;
* Any significant psychiatric disease;
* Use of illicit drugs;
* Unstable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate standing or stepping;
* Painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or urinary tract infection that might interfere with stand or step training;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Motor changes (MRC) | Before surgery, then monthly up to 6-month from surgery
  The Medical Research Council's (MRC) scale of muscle power will be used to evaluate motor weakness. The MRC scale of muscle strength uses a score from Grade 5 (normal) to Grade 0 (no visible contraction) to assess the power of a particular muscle group in relation to the movement of a single joint.
Motor changes (LEFS)) | Before surgery, then monthly up to 6-month from surgery
  The Lower Extremity Functional Scale (LEFS) will be used by clinicians as a measure of lower extremity function. It is a questionnaire containing 20 questions about a person's ability to perform everyday tasks (minimum score 0, maximum score 80).

SECONDARY OUTCOMES:
Spasticity changes | Before surgery, then monthly up to 6-month from surgery
  The Modified Ashworth scale will be used to evaluate spasticity. This scale grades the muscle tone from 0 (normal) to 4 (severe spasticity).
Longitudinal neurophysiological reorganization (electromyography) | Before surgery and 6 months after procedure
  Electromyography will be used to evaluate muscle response or electrical activity in response to a nerve's stimulation.
Longitudinal neurophysiological reorganization (motor evoked potentials) | Before surgery and 6 months after procedure
  Motor evoked potentials will be used to evaluate electrical signals recorded from the descending motor pathways or from muscles following stimulation of motor pathways within the brain.
Longitudinal neurophysiological reorganization (sensory evoked potentials) | Before surgery and 6 months after procedure
  Sensory evoked potentials will be used to assess electrical activity in the brain in response to sensory stimulation.
Longitudinal brain and spine MRI reorganization | Before surgery and 6 months after procedure
  Structural and functional brain and spine MRI analysis.
Chronic pain changes (MPQ) | Before surgery and 6 months after procedure
  The McGill Pain Questionnaire (MPQ) can be used to evaluate a person experiencing significant pain. It consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Chronic pain changes (PCS) | Before surgery and 6 months after procedure
  The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking. It assesses the extent of catastrophic thinking due to low back pain according to 3 components: rumination, magnification, and helplessness. It is a 13-item scale, with a total range of 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.
Chronic pain changes (ASC-12) | Before surgery and 6 months after procedure
  12-item Allodynia Symptom Checklist (ASC-12) evaluates presence of allodynia and hypoesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jackson A, Zimmermann JB. Neural interfaces for the brain and spinal cord--restoring motor function. Nat Rev Neurol. 2012 Dec;8(12):690-9. doi: 10.1038/nrneurol.2012.219. Epub 2012 Nov 13. PMID 23147846
- [Result] Sdrulla AD, Guan Y, Raja SN. Spinal Cord Stimulation: Clinical Efficacy and Potential Mechanisms. Pain Pract. 2018 Nov;18(8):1048-1067. doi: 10.1111/papr.12692. Epub 2018 Apr 23. PMID 29526043
- [Result] Seanez I, Capogrosso M. Motor improvements enabled by spinal cord stimulation combined with physical training after spinal cord injury: review of experimental evidence in animals and humans. Bioelectron Med. 2021 Oct 28;7(1):16. doi: 10.1186/s42234-021-00077-5. PMID 34706778
- [Result] Gill ML, Grahn PJ, Calvert JS, Linde MB, Lavrov IA, Strommen JA, Beck LA, Sayenko DG, Van Straaten MG, Drubach DI, Veith DD, Thoreson AR, Lopez C, Gerasimenko YP, Edgerton VR, Lee KH, Zhao KD. Neuromodulation of lumbosacral spinal networks enables independent stepping after complete paraplegia. Nat Med. 2018 Nov;24(11):1677-1682. doi: 10.1038/s41591-018-0175-7. Epub 2018 Sep 24. PMID 30250140
- [Result] Angeli CA, Boakye M, Morton RA, Vogt J, Benton K, Chen Y, Ferreira CK, Harkema SJ. Recovery of Over-Ground Walking after Chronic Motor Complete Spinal Cord Injury. N Engl J Med. 2018 Sep 27;379(13):1244-1250. doi: 10.1056/NEJMoa1803588. Epub 2018 Sep 24. PMID 30247091
- [Result] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197